CLINICAL TRIAL: NCT03255070
Title: A Phase 1, Multicenter, Open-label, Multiple Dose-escalation and Expansion Study of ARX788, as Monotherapy in Advanced Solid Tumors With HER2 Expression
Brief Title: A Dose-escalation, Expansion Study of ARX788, in Advanced Solid Tumors Subjects With HER2 Expression (ACE-Pan Tumor 01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ambrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARX788-1711
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Breast Neoplasms; Gastric Neoplasm; Solid Tumors
Keywords: HER2; antibody drug conjugate; breast cancer; gastric cancer; advanced solid tumors; HER2-overexpression; HER2-mutations
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — ARX788; Immunoconjugates

STUDY DESIGN:
Intervention Model Description: This is a 2-part, Phase 1, open-label study will administer the IMP, ARX788 by IV infusion every 3, 4 or 6 weeks. Sequential dose escalation cohorts are planned using a 3+3 design. A cohort may be expanded to collect additional data if recommended by Safety Monitoring Committee based on comprehensive reviews of safety, tolerability and PK data to determine RP2D.
  Phase 1a will determine the recommended Phase 2 dose (RP2D) in subjects with advanced cancer whose HER2 test results are in situ hybridization (ISH) positive or immunohistochemistry (IHC) 3+.
  Phase 1b will assess anticancer activity and safety in advanced cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARX788 Phase 1a (Dose Escalation) (Experimental): ARX788 will be administered every 3 weeks (Q3W) or every 4 weeks (Q4W) via intravenous (IV) infusion. Patients will be enrolled into escalating dose levels during Dose Escalation period.
  Interventions: Drug: ARX788
- ARX788 Phase 1b (Dose Expansion) (Experimental): ARX788 will be administered every 3 weeks (Q3W) via intravenous (IV) infusion. Patients will receive the maximum tolerated dose during the Dose Expansion period of the study.
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — An antibody drug conjugate
  Other Names: antibody drug conjugate (ADC)

SUMMARY:
This 2-part, Phase 1, open-label study will determine the recommended Phase 2 dose (RP2D) of ARX788 in subjects with advanced HER2 positive cancers and will assess the safety and anticancer activity in breast, gastric and other advanced HER2 positive solid tumors.

DETAILED DESCRIPTION:
Phase 1a will determine the recommended Phase 2 dose (RP2D) in subjects with advanced cancer whose HER2 test results are in situ hybridization (ISH) positive or immunohistochemistry (IHC) 3+, based on safety, tolerability, PK findings and antitumor activity. Phase 1b will assess the safety, tolerability, and PK and anticancer activity in five expansion cohorts, including breast cancer, gastric cancer / gastroesophageal adenocarcinoma, and other advanced HER2-positive solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Life expectancy >3 months.
* Female or male subjects whose advanced HER2 expressing cancer has failed standard of care treatments, or for whom such therapy is not acceptable to the subject. Subjects with advanced breast, gastric cancer, or other solid tumor who test positive for HER2 by ASCO/CAP criteria (either IHC or FISH) must have received prior treatment with a trastuzumab containing therapy. Subjects who have been previously treated with pertuzumab, TDM-1, lapatinib, or other available and accessible HER2-directed therapies or investigational therapies are eligible.
* Disease measurability:

  * Phase 1a: measurable or non-measurable disease per RECIST v 1.1.
  * Phase 1b: measurable disease per RECIST v 1.1 (subjects with non-measurable disease are not eligible for Phase 1b).
* Histopathologic evidence of cancer based upon pathology report.
* Tumor tissue local laboratory HER2 testing results, adequate tumor sample available for confirmation of HER2 status. Subjects with other types of cancer must have previously tested locally for HER2 status by HER2 IHC or ISH assay.

  * Phase 1a: ISH positive or IHC 3+ advanced cancer (including breast or gastric/esophageal or other solid tumors).
  * Phase 1b: Cohort 8 advanced breast cancer (IHC 3+ or IHC 2+/ISH); Cohort 9 advanced breast cancer (IHC 2+ / ISH-); Cohort 10 advanced gastric cancer (IHC 3+ or IHC 2+/ISH+) or gastroesophageal junction adenocarcinoma; Cohort 11 other advanced solid tumor cancers with HER2-overexpression (HER2 IHC 3+ or IHC 2+/IHS+); Cohort 12 advanced solid tumor cancers with HER2 activating mutation.
* Eastern Cooperative Oncology Group Performance Status of 0 to 1.
* Acute toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade 0 or 1 as per the NCI-CTCAE v 4.03 (phase 1a) and v 5.0 ( Phase 1b).
* Adequate organ functions.
* Willing and able to understand and sign an informed consent inform and to comply with all aspects of the protocol.
* Female subjects must be surgically sterile, or have a monogamous partner who is surgically sterile, or at least 2 years postmenopausal, or who commits to use an acceptable form of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence) for the duration of the study and for 3 months following the last dose of study treatment.
* Male subjects must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study.

Exclusion Criteria:

* History of allergic reactions to any component of ARX788.
* History of ocular events, or any current ongoing active ocular infections.
* History of congestive heart failure, unstable angina pectoris, unstable atrial fibrillation, or cardiac arrhythmia within 12 months prior to enrollment
* Grade 2 to 4 peripheral neuropathy (NCI CTCAE v 5.0)
* History of unstable central nervous system (CNS) metastases
* Current severe, uncontrolled systemic disease (eg, clinical significant cardiovascular, pulmonary, or metabolic diseases)
* Any uncontrollable intercurrent illness, infection (including subjects with active, symptomatic Covid-19 infections), or other conditions that could limit study compliance or interfere with assessments.
* Exposure to any other investigational or commercial anticancer agents or therapies administered with the intention to treat malignancy within 14 days before the first dose of ARX788.
* Clinically significant surgical intervention (excluding diagnostic biopsy) within 21 days of the first dose of ARX788
* Radiotherapy administered less than 21 days prior to the first dose of ARX788, or localized palliative radiotherapy administered less than 7 days prior to the first dose of ARX788, or radiotherapy-induced toxicity of Grade 2 or greater based on NCI-CTCAE v 5.0.
* Pregnancy or breast feeding.
* Known active HCV, HBV, and/or HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events, frequency and seriousness of treatment emergent adverse events (TEAEs) | Day 1 through 30 days after last dose
  To assess the safety, tolerability, and immunogenicity profile
Phase 1b: Objective response rate (ORR: complete response + partial response) per imaging assessment based on RECIST version 1.1. | 36 months
  Number of subjects with objective response is assessed every 6-8 weeks from Cycle 1 Day 1 through disease progression.

SECONDARY OUTCOMES:
Number of subjects with tumor response per imaging assessment based on RECIST version 1.1. | 18 months
  The objective response rate (ORR: CR+PR) based on RECIST v1.1 will be assessed as the primary endpoint to determine the anticancer activity of ARX788 as well as best overall response.
Area under the concentration-time curve (AUC) from first infusion to subject end of study. | 36 months
  Pharmacokinetic (PK) characteristics: ARX788 (intact ADC), total mAb, and metabolites
Half-life of ARX788 from first infusion to end of study. | 36 months
  Pharmacokinetic (PK) characteristics: ARX788 from first infusion to subject end of study
Immunogenicity profile of ARX788 | 36 months
  Number of subjects who develop anti-ARX788 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Ambrx, Study Director — Ambrx, Inc.
Locations (12):
- United States (5):
  - USC Norris Cancer Hospital, Los Angeles, California
  - UCLA Hematology-Oncology, Santa Monica, California
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor Sammons Cancer Center, Dallas, Texas
- Australia (7):
  - Research Site, East Albury, New South Wales
  - Research Site, North Sydney, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Princess Alexandria Hospital, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - Research Site, Frankston, Victoria
  - Research Site, Nedlands, Western Australia